CLINICAL TRIAL: NCT00671489
Title: Phase 2 Study of Tachikawa Project for Prevention of Posttraumatic Stress Disorder With Polyunsaturated Fatty Acid (TPOP): TPOP-01 Study
Brief Title: Tachikawa Project for Prevention of Posttraumatic Stress Disorder With Polyunsaturated Fatty Acid (TPOP): TPOP-01 Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Japan Science and Technology Agency (Other)
Collaborators: University of Toyama (Other); Chiba University (Other)
Responsible Party: Matsuoka Yutaka, National Disaster Medical Center and National Center of Neurology and Psychiatry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NDMC-TPOP-01
Record Dates: First submitted 2008-04-23; First posted 2008-05-05 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2009-05

CONDITIONS: Trauma; Posttraumatic Stress Disorder
Keywords: Patients; high-energy; admitted; intensive care unit; motor vehicle accident; falling from height; other accident
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Omega-3 Polyunsaturated Fatty Acid — A capsule of omega-3 Polyunsaturated Fatty Acid, 300mg (including 70% docosahexaenoic acid, 7% eicosapentaenoic acid and other), 7 capsules per day in 12 week.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Polyunsaturated Fatty Acid for the prevention of Posttraumatic Stress Disorder (PTSD) in patients with accidental injuries.

DETAILED DESCRIPTION:
Accidental injuries, mostly motor vehicle accident, in civilian population are frequent events. For instance, nearly one-third of injured patients appear to develop trauma-related psychiatric illness and the major diagnoses are post-traumatic stress disorder (PTSD) and depressive disorder. Omega-3 Polyunsaturated Fatty Acid (Omega-3 PUFA) has some evidence of efficacy of treatment in patients with anxiety and mood disorders, but no evidence of preventing anxiety and mood disorders that occur subsequent to accidental injuries. We evaluate efficacy and safety of Omega-3 PUFA for the secondary prevention of Posttraumatic Stress Disorder (PTSD) and related psychiatric illness in patients with accidental injury.

ELIGIBILITY:
Inclusion Criteria:

1. 18 plus years
2. A native Japanese speaking ability
3. Possibility contact patients with injury in 240 hours, and dosing in oral use
4. Physical and metal status to possible understands scope and contents in the trial and gets informed consent

Exclusion Criteria:

1. Clearly irretrievable acute brain parenchyma damage and subdural or subarachnoidal bleeding detected by computed tomography and/or magnetic resonance imaging
2. Cognitive impairment: Mini Mental State Examination < 24
3. Heavy drinker or 100IU/L ≦ γGTP in administration
4. Heavy smoker (over 40 cigarettes per day)
5. History and current suspicion in diagnosis of psychosis and bipolar I disorder
6. Suspicion in diagnosis of alcoholic, substance-related disorder and eating disorder
7. Existence of marked serious symptoms such as suicidal ideation, self-harm behavior, dissociation, status of need rapidly psychiatric treatment
8. Use of anti-epilepsy drug, lithium, ethyl icosapentate and anti-coagulant drug (for example, aspirin, warfarin, etc) within 3 month at regular intervals
9. Use of polyunsaturated fatty acid supplement within 3 month at regular intervals
10. Habit of eating fish over 4 times per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Total score of Clinician-Administrated PTSD Scale (CAPS) | Three month

SECONDARY OUTCOMES:
Incidence of diagnosis of PTSD (including partial PTSD) | Three month, one month
Total score of Montgomery Asberg Depression Rating Scale (MADRAS) | Three month, one month
Incidence of depression evaluated by Mini-International Neuropsychiatric Interview (MINI) | Three month, one month
Autonomic response measured before, during and after script driven imagery and acoustic stimulation | Three month
Score of Impact of Event Scale revised (IES-R) | Three month, one month
Score of Hospital Anxiety and Depression scale (HADS) | Three month, one month
Score of health related Quality of Life scale, SF-36 | Three month, one month
Score of Conner-Davidson Resilience Scale (CD-RISC) | Three month, one month
Brain-derived neurotrophic factor (BDNF) in serum | Three month, one month
Number of days of leave taken from the time of injury | Three month
Buss-Perry Aggression Questionnaire (BAQ) | Three month, one month, baseline
Total score of Clinician-Administrated PTSD Scale (CAPS) | One month
DHEA: dehydroepiandrosterone | Three month, one month
NPY: neuropeptide Y | Three month, one month
IL-1 beta: interleukin 1 beta | Three month, one month
IL-6: interleukin 6 | Three month, one month
TNF alpha: tumor necrosis factor alpha | Three month, one month
D-serine | Three month, one month
L-serine | Three month, one month
DL-serine | Three month, one month
Activin | Three month, one month

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Mastuoka, M.D., Ph.D., Principal Investigator — National Disaster Medical Center, Tachikawa, Tokyo ,Japan
Locations (1):
- National Disaster Medical Center, Tachikawa, Tokyo ,Japan, Tachikawa, Tokyo, Japan

REFERENCES:
- [Result] Matsuoka Y, Nishi D, Yonemoto N, Hamazaki K, Hashimoto K, Hamazaki T. Omega-3 fatty acids for secondary prevention of posttraumatic stress disorder after accidental injury: an open-label pilot study. J Clin Psychopharmacol. 2010 Apr;30(2):217-9. doi: 10.1097/JCP.0b013e3181d48830. No abstract available. PMID 20520307
- [Result] Matsuoka Y. Clearance of fear memory from the hippocampus through neurogenesis by omega-3 fatty acids: a novel preventive strategy for posttraumatic stress disorder? Biopsychosoc Med. 2011 Feb 8;5:3. doi: 10.1186/1751-0759-5-3. PMID 21303552
- [Result] Matsuoka Y, Nishi D, Yonemoto N, Hamazaki K, Hamazaki T, Hashimoto K. Potential role of brain-derived neurotrophic factor in omega-3 Fatty Acid supplementation to prevent posttraumatic distress after accidental injury: an open-label pilot study. Psychother Psychosom. 2011;80(5):310-2. doi: 10.1159/000322980. Epub 2011 Jun 30. No abstract available. PMID 21720194